CLINICAL TRIAL: NCT01089660
Title: Immunogenicity of the Intramuscular Inactivated, Split Virion Swine-origin A/H1N1 Influenza Vaccine Without Adjuvant in Healthy Adult Subjects
Brief Title: A Study of the Immunogenicity of Swine-origin A/H1N1 Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GPF18; 2010-018991-25 (EudraCT Number); UTN: U1111-1112-8378 (Other: WHO)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza; Pandemic Flu; Swine-origin Influenza; Inactivated split-virion vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group 1 (Experimental): Swine-origin A/H1N1 Vaccine Low-dose
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)
- Study Group 2 (Experimental): Swine-origin A/H1N1 Vaccine High-dose
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)

INTERVENTIONS:
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.3 mL, Intramuscular (IM)
  Arms: Study Group 1
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.5 mL, Intramuscular (IM)
  Arms: Study Group 2

SUMMARY:
This study is designed to describe the immunogenicity of a pandemic A/H1N1 influenza vaccine in healthy adults given a lower vaccine dose and in a similar group given a full dose of the vaccine.

The primary objective is to describe describe the immune response of the inactivated, split-virion swine-origin A/H1N1 influenza vaccine without adjuvant.

DETAILED DESCRIPTION:
All participants will receive a single dose of study vaccine and will also be monitored for serious adverse events and adverse events of special interest occurring from Days 0 to 21 and at 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 60 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination
* Entitled to national social security

Exclusion Criteria :

* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator
* Participant previously vaccinated with an A/H1N1 pandemic influenza vaccine during vaccination campaign or in a clinical trial
* Personal history of influenza infection since May 2009
* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity in terms of anti-hemagglutinin (HA) antibody titers against non-adjuvanted pandemic A/H1N1 influenza vaccine. | 21 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- France (2):
  - Rennes
  - Rueil-Malmaison

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com